CLINICAL TRIAL: NCT01274494
Title: COMPLIANCE An Observational Study of Treatment Compliance and Quality of Life in Patients on Antihypertensive Medication
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CME-ATA-2010/1
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: High Blood Pressure
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this multi-centre survey is to assess treatment adherence and quality of life in a Jordanian and Lebanese population newly diagnosed with hypertension or with uncontrolled essential hypertension being on antihypertensive treatment for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 21 years of age
* Patients newly diagnosis with essential hypertension or with hypertension that is uncontrolled after being under the same antihypertensive treatment for at least 6 months (based on the criteria established by the Joint National Committee VII)
* Patients capable of providing an informed consent

Exclusion Criteria:

* Patients with secondary hypertension
* Pregnant women or nursing mothers
* Patients with acute illnesses or psychiatric diagnosis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multi-centre survey of patients
Sampling Method: Non-Probability Sample
Enrollment: 1501 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Compliance rate | 6 months
  Identify the percentage of subjects compliant to their antihypertensive treatment.

SECONDARY OUTCOMES:
Health Related Quality of Life (MINICHAL Score) | 6 months
  To compare and identify changes in the quality of life before and after anti-hypertensive treatment.
Type of pharmacological treatments | 6 months
  To identify the pharmacological treatments used by physicians in Jordan and Lebanon to treat patients newly diagnosed or with uncontrolled hypertension.
Factors affecting adherence to treatment | 6 months
  To identify associated factors that may alter adherence to anti-hypertensive treatment.
Compliance rate by antihypertensive regimen used | 6 months
  To compare treatment rate for different antihypertensive regimen used
Percentage of controlled patients | 6 months
  To identify the percentage of patients reaching their target blood pressure according to the JNCVII criteria.